CLINICAL TRIAL: NCT06104176
Title: Effectiveness of Virtual Reality Therapy in Alcohol Use Disorder Study : a Multicenter Randomized Trial. Original Title in French : étude de l'efficacité de la Réalité Virtuelle Dans le Traitement du Trouble de l'Usage d'Alcool : un Essai randomisé Multicentrique (e-Réva)
Brief Title: Effectiveness of Virtual Reality Therapy in Alcohol Use Disorder Study
Acronym: e-ReVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP221352
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Alcool Use Disorder
MeSH Terms: interventions — Population Groups; Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT group (Active Comparator)
  Interventions: Behavioral: CBT in group; Behavioral: individual CBT
- VRET group (Experimental)
  Interventions: Behavioral: CBT in group; Other: Virtual reality exposure

INTERVENTIONS:
Behavioral: CBT in group — All subjects will have 4 sessions of group CBT (one per week) during the first month following their inclusion, and then randomly assigned (ratio 1:1) to VRET group or individual CBT group. Subjects will undergo 4 additional sessions of VRET or individual CBT (one per week) during the second month.
  VRET consists on 4 weekly sessions (one per week, for 1 month) of 60 to 90 minutes duration. Each session, consists in 20 to 30 minutes exposure with 10 minutes breaks (2 to 3 exposure per session). Four environments will be used: The home environment, the metro advertising environment , the party environment, and the supermarket environment. Each session corresponds to one environment, previously ordered according to their difficulty for the patient.
Other: Virtual reality exposure — ll subjects will have 4 sessions of group CBT (one per week) during the first month following their inclusion, and then randomly assigned (ratio 1:1) to VRET group or individual CBT group. Subjects will undergo 4 additional sessions of VRET or individual CBT (one per week) during the second month.
  VRET consists on 4 weekly sessions (one per week, for 1 month) of 60 to 90 minutes duration. Each session, consists in 20 to 30 minutes exposure with 10 minutes breaks (2 to 3 exposure per session). Four environments will be used: The home environment, the metro advertising environment , the party environment, and the supermarket environment. Each session corresponds to one environment, previously ordered according to their difficulty for the patient.
  Arms: VRET group
Behavioral: individual CBT — ll subjects will have 4 sessions of group CBT (one per week) during the first month following their inclusion, and then randomly assigned (ratio 1:1) to VRET group or individual CBT group. Subjects will undergo 4 additional sessions of VRET or individual CBT (one per week) during the second month.
  VRET consists on 4 weekly sessions (one per week, for 1 month) of 60 to 90 minutes duration. Each session, consists in 20 to 30 minutes exposure with 10 minutes breaks (2 to 3 exposure per session). Four environments will be used: The home environment, the metro advertising environment , the party environment, and the supermarket environment. Each session corresponds to one environment, previously ordered according to their difficulty for the patient.
  Arms: CBT group

SUMMARY:
Intro: Virtual reality exposure therapy (VRET) has been widely assessed in several mental disorders, including substances use disorders. In the case of alcohol use disorder (AUD), published studies focus mainly on craving interventions: eliciting, triggering, reduction or extinction, with promising result. However, data Virtual reality exposure therapy effect on reduction of alcohol consumption or abstinence remains scarce.

Hypothesis/Objective: The investigators hypothesis that VRET associated to cognitive behaviors therapy (CBT) will be more effective than CBT alone on the reduction in the cumulative number of standard drinks (vs) of alcohol intakes at 8 months after inclusion. The second objective is the assess its effectiveness on reported craving also at 8 months.

Method: The investigators plane to recruit 156 subjects aged 18 and over, with AUD according to DSM V criteria, abstinent for at least 15 days. Non-inclusion criteria are: AUD relapse, pregnancy or breastfeeding (for women), decompensated comorbid mental disorder, severe cognitive impairment, epilepsy or history of photo paroxysmal EEG responses, balance disorders, recent stroke less than 3 months old, current nausea/vomiting, claustrophobia, severe visual impairment, and medium or high myopia (beyond -3.5 diopters). The study recruitment and sitting will be on 4 addiction day hospitals, and the follow up period will be of 8 months.

All subjects will have 4 sessions of group CBT (one per week) during the first month following their inclusion, and then randomly assigned (ratio 1:1) to VRET group or individual CBT group. Subjects will undergo 4 additional sessions of VRET or individual CBT (one per week) during the second month. Afterwards, all included subjects will be followed monthly for 6 months (Months 2 to 8 after inclusion). Timeline Follow-Back (TLFB) is used for the reporting of the number of alcohol standard drinks intakes, and the Transaddiction Craving Triggers Questionnaire (TCTQ) for craving assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over, and under 80 on the date of inclusion
* Fulfilling Alcohol use disorder according to the DSM-V criteria (American Psychiatric Association, 2013);
* In alcohol abstinence for at least 15 days;
* Be able to speak, understand and read French;
* Signed an informed consent
* Affiliated to the French health insurance scheme

Exclusion Criteria:

* • Major under legal protection measure, or deprived of liberty by judicial or administrative decision;

  * Pregnant or breastfeeding women;
  * Decompensated psychiatric disoreder (psychotic disorders, mood disorders and anxiety disorders);
  * Alcohol use disorder relapse
  * Severe cognitive impairment as defined by a score of 10 or less at the Montreal Cognitive Assessment (MOCA) (Nasreddine et al., 2005)
  * Visual impairment
  * Contraindications to virtual reality exposure: a history of photosensitive epilepsy, response, balance disorders, recent stroke less than 3 months old, current nausea/vomiting, claustrophobia, and medium or high myopia (beyond -3.5 diopters)
  * Patients wearing one of the following medical devices (due to the risk of interference of the virtual reality headset with them): pacemaker, implanted defibrillator, or implanted hearing aids (non-implanted prostheses are not contraindicated if the patient agrees to remove them during virtual reality exposure)
  * Participation in another trial or being in the exclusion period following previous research involving humans, if applicable
  * Patients not affiliated to the French health insurance scheme and receiving the State Medical Aid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative number of alcohol standard drinks | monthly until 8 months after inclusion
  Cumulative number of alcohol standard drinks 8 months after inclusion assessed by the Timeline Follow-Back method (Sobell & Sobell, 1992).

SECONDARY OUTCOMES:
Craving | at inclusion, 2, 5 and 8 months after inclusion
  Level of reported craving assessed by the Transaddiction Craving Triggers Questionnaire (von Hammerstein et al., 2020) and by a Visual Analogue Scale (from 0 to 10) (Drobes & Thomas, 1999).
frequency of alcohol hazardous drinks | at inclusion, 2, 5 and 8 months after inclusion
  the frequency is assessed by the Alcohol Use Disorders Identification Test (AUDIT-C) (Bush et al., 1998)
Anxiety level | at inclusion, 2, 5 and 8 months after inclusion
  Anxiety level is assessed by the (Generalized Anxiety Disorder-7) (Spitzer et al., 2006)
Depression severity | at inclusion, 2, 5 and 8 months after inclusion
  Depression symptoms severity are assessed by the Patient Health Questionnaire 9) (Kroenke et al., 2001).
Self-efficacy | at inclusion, 2, 5 and 8 months after inclusion
  Self-efficacy is assessed by Self-efficacy Questionnaire (Jerusalem & Schwarzer, 1992).
Repetitive thinking | at inclusion, 2, 5 and 8 months after inclusion
  Repetitive negative thinking is assessed by the The Perseverative Thinking Questionnaire (PTQ) en (Devynck et al, 2017)
Virtual environment presence | at inclusion, 2, 5 and 8 months after inclusion
  Virtual environment presence is assessed by the presence questionnaire (Witmer et al.2005)
Cybersickness | at inclusion, 2, 5 and 8 months after inclusion
  Cybersickness symptoms are assessed by the Simulator Sickness Questionnaire (Kennedy et al., 1993)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Albert Chenevier, Créteil, Île-de-France Region, France

REFERENCES:
- [Derived] Negre F, Lemercier-Dugarin M, Gomet R, Pelissolo A, Malbos E, Romo L, Zerdazi EH. Study on the efficiency of virtual reality in the treatment of alcohol use disorder: study protocol for a randomized controlled trial : E-Reva. Trials. 2024 Jun 27;25(1):417. doi: 10.1186/s13063-024-08271-x. PMID 38937776